CLINICAL TRIAL: NCT05222438
Title: Phase II Trial Evaluating Safety and Efficacy of Loncastuximab Tesirine as a Maintenance Therapy Following Autologous Stem Cell Transplantation in High Risk Diffuse Large B-cell Lymphoma
Brief Title: Trial of Loncastuximab Tesirine in High Risk Diffuse Large B-cell Lymphoma Post Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No accrual of participants in 18 months
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Dipenkumar Modi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-047; ADCT-402-001 (Other: ADC Therapeutics)
Record Dates: First submitted 2022-01-10; First posted 2022-02-03 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Relapsed Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Loncastuximab tesirine (Experimental): Patients will start loncastuximab tesirine for maintenance therapy between day 30 and 60 following autoSCT and will receive a total of 6 months of therapy (8 cycles). Patients will receive IV infusion of loncastuximab tesirine 150 μg/kg at Q3W for the first 2 cycles followed by 75 μg/kg at Q3W for the remaining 6 cycles.
  Interventions: Drug: loncastuximab tesirine

INTERVENTIONS:
Drug: loncastuximab tesirine — loncastuximab tesirine for maintenance therapy between day 30 and 60 following autoSCT and will receive a total of 6 months of therapy (8 cycles).

SUMMARY:
Study of loncastuximab tesirine administered intravenously (IV) for maintenance therapy following autologous stem cell transplant in patients with relapsed diffuse large B cell lymphoma

DETAILED DESCRIPTION:
This is a Phase II, multicenter, open label study of loncastuximab tesirine for maintenance therapy following autologous stem cell transplant (autoSCT) in patients with relapsed diffuse large B cell lymphoma (DLBCL). Patients with relapsed DLBCL confirmed through core biopsy and meeting eligibility criteria will be enrolled in the study. Patients can be enrolled up to 4 weeks prior to autoSCT. Patients will start loncastuximab tesirine between day 30 and 60 after autoSCT as determined by the treating physician. Since majority of the relapses occur early after autoSCT, offering maintenance therapy for a finite duration might be of therapeutic benefit without posing excessive toxicity. Loncastuximab tesirine will be administered intravenously (IV) at every 3 weeks (Q3W) for a total of 6 months (8 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF)
2. Age >18 years
3. Patients with relapsed refractory DLBCL with any of the following high-risk features for progression following autoSCT will be enrolled:

   * Primary refractory lymphoma (failure to achieve complete remission as determined by the treating physician) following 1st line anthracycline containing chemotherapy
   * Early relapsed lymphoma with an initial remission duration of less than 12 months following 1st line anthracycline containing chemotherapy
   * Failure to achieve complete remission following salvage chemotherapy and positive PET-CT as defined by Lugano criteria (Deauville score of 4 or 5) prior to autoSCT
   * Double hit lymphoma (DHL) or triple hit lymphoma (THL) confirmed by FISH testing by local pathology (defined as high grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements)
   * Double expressor lymphoma (DEL) as confirmed by immunohistochemistry (IHC) by local pathology (MYC and BCL2 or BCL6 positivity)
   * CMYC rearranged (by FISH) DLBCL
   * High IPI score (≥3 points)
   * Stage 3-4 disease at diagnosis
   * Extra-lymphatic disease
   * High grade B cell lymphoma
4. Eligible to undergo autologous stem cell transplantation as per local investigator assessment
5. Availability of biopsy specimens confirming DLBCL relapse. Archival formalin-fixed paraffin-embedded (FFPE) tissue blocks or 15 unstained slides serial sections (5-10 μm in thickness) must be available prior to study enrollment. The pathology report must be available. IHC testing of CMYC, BCL2, and BCL6 expression, and FISH testing of CMYC, BCL2 and BCL6 gene rearrangement must be available prior to enrollment. CD19 expression status must be available prior to enrollment.
6. Patients previously treated with CD19-targeted therapy (including CAR T) must have a subsequent biopsy and/or flow cytometry confirming CD19 positivity.
7. ECOG Performance Status of 0, 1, or 2
8. Life expectancy of at least 6 months
9. Ability and willingness to comply with the study protocol procedures
10. Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 9 months after the last dose of loncastuximab tesirine. Men with female partners who are of childbearing potential must agree that they will use a highly effective method of contraception from the time of giving informed consent until at least 6 months after the patient receives his last dose of loncastuximab tesirine

Exclusion Criteria:

1. Contraindications to any of the individual components of autoSCT or loncastuximab tesirine.
2. Prior exposure to loncastuximab tesirine
3. Clinically significant effusion i.e. ascites, pleural or pericardial effusion requiring drainage or associated with shortness of breath
4. Patients with ongoing toxicities of grade >1 from previous treatments except alopecia
5. Patients with clinically significant history of liver disease including cirrhosis or hepatitis (viral hepatitis). However, treated viral hepatitis may be allowed Patients with history of severe skin disorders including Steven-Johnson syndrome (SJS) or toxic epidermal necrolysis (TEN)
6. Patients who are receiving any other investigational agents
7. Grade 3b follicular lymphoma
8. Burkitt's lymphoma
9. Patients with known brain, spinal, or CSF involvement
10. Systemic steroids (prednisone >20 mg/day or equivalent) and/or immunosuppressive medications
11. Unstable cardiovascular function that could affect compliance with the protocol:

    * Symptomatic ischemia, or
    * Congestive heart failure (CHF) of NYHA Class ≥3, or
    * Myocardial infarction (MI) within 3 months
    * Left ventricular ejection fraction <45% based on echocardiogram or MUGA scan obtained within 6 months prior to enrollment
    * History or presence of an abnormal ECG that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block.
12. Positive test results for chronic hepatitis B virus (HBV) infection (defined as positive hepatitis B surface antigen [HBsAg]):

    -Patients with occult or prior HBV infection (defined as negative HBsAg and positive hepatitis B core antibody [HBcAb]) may be included if HBV DNA PCR is undetectable, provided that they are willing to undergo DNA testing on Day 1 of every cycle of study treatment. Patients who have protective titers of hepatitis B surface antibody (HBsAb) after vaccination or prior but cured hepatitis B are eligible.
13. Known history of HIV seropositive status
14. Patients with a history of progressive multifocal leukoencephalopathy
15. Any of the following, unless abnormal laboratory values are due to underlying lymphoma per the investigator:

    * Creatinine > 1.5 x ULN or a measured creatinine clearance < 40 mL/min
    * AST or ALT > 2.5 x ULN
    * Total bilirubin > 1.5 x ULN. Patients with documented Gilbert disease may be enrolled if total bilirubin is < 3 x ULN
    * INR or PT > 1.5 x ULN in the absence of therapeutic anticoagulation
    * PTT or aPTT > 1.5 x ULN in the absence of a lupus anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-08 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy Outcome Measure | From the start date of treatment initation until the date of progression or death from any cause, whichever occurs first, assessed up to 1-year following autoSCT
  Progression-free survival (PFS) assessments will be determined according to Lugano Response Criteria. The distributions of time to event data will be graphically summarized using Kaplan-Meier (KM) curves and their median and confidence intervals will be estimated using KM estimates.
Safety Outcome Measure | Up to 30 days after last dose of study treatment
  Evaluate the safety and tolerability as defined by CTCAE 5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Dipenkumar Modi, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States